CLINICAL TRIAL: NCT03567070
Title: Pregnancy and Use of Psychoactive Substances: The Influence of Representations of Care on Care.
Acronym: ADDGEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-050
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- qualitative study based on an individual clinical interview (Other)
  Interventions: Other: qualitative study based on an individual clinical interview

INTERVENTIONS:
Other: qualitative study based on an individual clinical interview — qualitative study based on an individual clinical interview

SUMMARY:
It is observed that pregnant women using psychoactive substance (s) have a more random and more accidental pregnancy follow-up than women with no addictive problems.

The consumption approach can be either omitted during the pregnancy monitoring, or entrusted to the course or more often in late pregnancy or occurs more brutally during delivery at the time of complications (neonatal or obstetric). In this context, health professionals are looking for levers that allow women to take appropriate care quickly.

This difficulty of access to care questions us and all the more because the time of the pregnancy is a moment of important psychic reorganization conducive to modify its habits, to change its glance on its consumptions and thus to start a care concerning addiction.

Invesigators hypothesize that this population has less access to medical care during pregnancy for fear of stigmatization by the health care provider.

Invesigators propose a multicenter qualitative study based on individual clinical interviews to collect the testimony of women who used psychoactive substance (s) during their pregnancy.

The purpose of this work is to identify ways to improve the multidisciplinary medical management of these women by focusing on the representations they can make care of.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Pregnant or having given birth since <28 days
* Having used (whether declared or discovered incidentally) - regardless of the amount of psychoactive substance (s) during pregnancy: alcohol, and / or heroin or OST, and / or cannabis, and / or psychostimulants (cocaine, ecstasy, amphetamines)
* Followed or not in addictology during pregnancy

Exclusion Criteria:

* Minor patients
* Patients under legal protection (guardianship, guardianship)
* Linguistic obstacle
* Psychiatric pathology decompensated at the time of the meeting
* Women who only used tobacco regularly during pregnancy
* Women who have only regularly used psychoactive drugs and / or licit opiates (excluding prescription replacement products) during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Enrollment: 9 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
individual clinical interview | baseline
  qualitative study based on an individual clinical interview

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No